CLINICAL TRIAL: NCT02094573
Title: A Randomized Phase 2 Study of AP26113 in Patients With ALK-positive, Non-small Cell Lung Cancer (NSCLC) Previously Treated With Crizotinib
Brief Title: A Study to Evaluate the Efficacy of Brigatinib (AP26113) in Participants With Anaplastic Lymphoma Kinase (ALK)-Positive, Non-small Cell Lung Cancer (NSCLC) Previously Treated With Crizotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP26113-13-201; 2013-002134-21 (EudraCT Number); U1111-1196-8246 (Other: WHO)
Record Dates: First submitted 2014-03-18; First posted 2014-03-24 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brigatinib 90 mg (Experimental): Brigatinib 90 mg, tablets, orally, once daily in each Cycle of 28 days until disease progression or intolerable toxicity (median duration of exposure was 402 days).
  Interventions: Drug: Brigatinib
- Brigatinib 90 mg - 180 mg (Experimental): Brigatinib 90 mg, tablets, orally, once daily for 7 days followed by brigatinib 180 mg, orally once daily in Cycle 1 of 28 days followed by brigatinib 180 mg, orally once daily in Cycle 2 and onward Cycles of 28 days until disease progression or intolerable toxicity (median duration of exposure was 522 days).
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib tablets
  Other Names: AP26113; ALUNBRIG™

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two different dosing regimens of brigatinib (AP26113) in participants with ALK-positive locally advanced or metastatic non-small cell lung cancer (NSCLC) whose disease has progressed on therapy with crizotinib.

DETAILED DESCRIPTION:
The drug being tested in this study is called brigatinib (AP26113). Brigatinib was tested to treat people with anaplastic lymphoma kinase (ALK)-positive metastatic non-small cell lung cancer (NSCLC) who have progressed on or were intolerant to crizotinib. This study looked at the efficacy of brigatinib.

The study enrolled 222 patients. Participants were randomly assigned (by chance, like flipping a coin) to one of the two treatment groups:

* Brigatinib 90 mg
* Brigatinib 90 mg -180 mg

All participants were asked to take a tablet, orally once daily until disease progression or intolerable toxicity. Participants in Brigatinib 90 mg - 180 mg received 180 mg with a 7-day lead-in at 90 mg.

This multi-center trial was conducted worldwide. The overall time to participate in this study is up to 3 years. Participants will make multiple visits to the clinic, and 3 months after the End-of-Treatment visit. Follow-up is intended to continue for 2 years after the last participants was enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) that is anaplastic lymphoma kinase (ALK+).
2. Must meet one of the following two criteria:

   1. Have documented ALK rearrangement by a positive result from the Vysis® ALK Break-Apart fluorescence in situ hybridization (FISH) Probe Kit; or
   2. Have documented ALK positivity by a different test and tissue available for the Vysis® FISH test. Tissue should be derived preferably from a biopsy taken after progression with crizotinib. If such a sample is not available, testing may be performed with archived tumor tissue.
3. Had progressive disease while on crizotinib, as assessed by the investigator or treating physician.
4. Have at least 1 measurable lesion per RECIST v1.1. Note: Previously irradiated lesions may not be used for target lesions, unless there is unambiguous radiological progression after radiotherapy. Brain lesions may not be used as target lesions if they were: 1) previously treated with whole brain radiation therapy (WBRT) within 3 months, or 2) previously treated by stereotactic radiosurgery (SRS) or surgical resection.
5. Recovered from toxicities related to prior anticancer therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE, v4.0) grade ≤2.
6. Are a male or female participants ≥18 years old.
7. Have a life expectancy ≥3 months.
8. Have adequate organ and hematologic function, as determined by:

   1. Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN; ≤5 x ULN is acceptable if liver metastases are present)
   2. Total serum bilirubin ≤1.5 x ULN (<3.0 x ULN for participants with Gilbert syndrome)
   3. Serum creatinine ≤1.5 x ULN
   4. Serum lipase/amylase ≤1.5 x ULN
   5. Absolute neutrophil count (ANC) ≥1500/µL
   6. Platelets ≥75000/µL
   7. Hemoglobin ≥10 g/dL
9. Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
10. Have normal QT interval on screening electrocardiogram (ECG) evaluation, defined as QT interval corrected (Fridericia) (QTcF) of ≤450 ms in males or ≤470 ms in females.
11. For female participants of childbearing potential, a negative pregnancy test must be documented prior to enrollment.
12. Female and male participants who are fertile must agree to use a highly effective form of contraception with their sexual partners throughout study participation.
13. Must provide a signed and dated informed consent indicating that the participants has been informed of all pertinent aspects of the study, including the potential risks, and is willingly participating.
14. Have the willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Received any prior ALK-targeted TKI other than crizotinib.
2. Received crizotinib within 3 days of the first dose of brigatinib (Day 1, Cycle 1).
3. Received cytotoxic chemotherapy, investigational agents, or radiation within 14 days, except SRS or stereotactic body radiosurgery.
4. Received monoclonal antibodies or had major surgery within 30 days of the first dose of brigatinib (Day 1, Cycle 1).
5. Have been diagnosed with another primary malignancy within the past 3 years (except for adequately treated non-melanoma skin cancer, cervical cancer in situ, or prostate cancer, which are allowed within 3 years).
6. Have symptomatic CNS metastases that are neurologically unstable or require an increasing dose of corticosteroids.
7. Have current spinal cord compression.
8. Have significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   1. Myocardial infarction (MI) within 6 months prior to the first dose of brigatinib
   2. Unstable angina within 6 months prior to first dose
   3. Congestive heart failure (CHF) within 6 months prior to first dose
   4. History of clinically significant (as determined by the treating physician) atrial arrhythmia
   5. Any history of ventricular arrhythmia
   6. Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose
9. Have a history or the presence of pulmonary interstitial disease or drug-related pneumonitis.
10. Have an ongoing or active infection. The requirement for intravenous (IV) antibiotics is considered active infection.
11. Have a known history of human immunodeficiency virus (HIV). Testing is not required in the absence of history.
12. Have a history of or active significant gastrointestinal (GI) bleeding within 3 months of the first dose of brigatinib.
13. Have a known or suspected hypersensitivity to brigatinib or its excipients.
14. Have malabsorption syndrome or other GI illness that could affect oral absorption of the study drug.
15. Have any condition or illness that, in the opinion of the investigator, would compromise participants safety or interfere with evaluation of the drug study.
16. Be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-06-04 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda

REFERENCES:
- [Derived] Kawata AK, Lenderking WR, Eseyin OR, Kerstein D, Huang J, Huang H, Zhang P, Lin HM. Converting EORTC QLQ-C30 scores to utility scores in the brigatinib ALTA study. J Med Econ. 2019 Sep;22(9):924-935. doi: 10.1080/13696998.2019.1624080. Epub 2019 Jun 25. PMID 31125274
- [Derived] Camidge DR, Kim DW, Tiseo M, Langer CJ, Ahn MJ, Shaw AT, Huber RM, Hochmair MJ, Lee DH, Bazhenova LA, Gold KA, Ou SI, West HL, Reichmann W, Haney J, Clackson T, Kerstein D, Gettinger SN. Exploratory Analysis of Brigatinib Activity in Patients With Anaplastic Lymphoma Kinase-Positive Non-Small-Cell Lung Cancer and Brain Metastases in Two Clinical Trials. J Clin Oncol. 2018 Sep 10;36(26):2693-2701. doi: 10.1200/JCO.2017.77.5841. Epub 2018 May 16. PMID 29768119

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 71 investigative sites in the United States, Canada, Europe, Australia, and Asia from 04 Jun 2014 to 27 February 2020.
Pre-assignment Details: Participants with diagnosis of anaplastic lymphoma kinase (ALK)-positive, non-small cell lung cancer (NSCLC) who had progressed on crizotinib were enrolled to receive brigatinib 90 mg, once daily or brigatinib 90-180 mg, once daily.
Period: Overall Study
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Started | 112 | 110
Treated | 109 | 110
Completed (Completed = Participants who completed the treatment.) | 0 | 0
Not Completed | 112 | 110
Not completed — Adverse Event | 4 | 14
Not completed — Clinical Progressive Disease | 9 | 13
Not completed — Death | 11 | 3
Not completed — Documented Progressive Disease (RECIST 1.1) | 63 | 50
Not completed — Non-compliance with Study Drug | 1 | 1
Not completed — Subject Received a New Systemic Anticancer Therapy | 1 | 0
Not completed — Physician Decision | 4 | 4
Not completed — Site Terminated by Sponsor | 10 | 17
Not completed — Withdrawal by Subject | 6 | 8
Not completed — Randomized but not Treated | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intention to Treat (ITT) Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhere to the assigned dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg | Total
Number analyzed (Participants) | 112 | 110 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.03) | 55.4 (12.98) | 53.4 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 64 | 126
  Male | 50 | 46 | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 72 | 76 | 148
  Black or African American | 1 | 2 | 3
  Asian | 39 | 30 | 69
  Unknown | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 107 | 102 | 209
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 6 | 9
  Austria | 3 | 6 | 9
  Belgium | 3 | 2 | 5
  Canada | 2 | 1 | 3
  Denmark | 2 | 6 | 8
  France | 4 | 2 | 6
  Germany | 7 | 7 | 14
  Hong Kong | 6 | 0 | 6
  Italy | 15 | 14 | 29
  Netherlands | 6 | 6 | 12
  Norway | 1 | 1 | 2
  Singapore | 4 | 3 | 7
  Spain | 5 | 7 | 12
  Sweden | 2 | 2 | 4
  Switzerland | 0 | 1 | 1
  United Kingdom | 2 | 1 | 3
  United States | 21 | 25 | 46
  Korea, Republic Of | 26 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR) as Assessed by Investigator
Description: ORR assessed by the investigator, was defined as percentage of the participants with confirmed complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST) v1.1 (confirmed ≥4 weeks after initial response), after initiation of study treatment. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline sum diameters. The exact 2-sided 97.5% confidence interval was calculated. The treatment regimen was considered to have achieved the primary objective when lower bound of the 97.5% confidence interval for ORR assessed by investigator is greater than 20%.
Time Frame: Screening, at 8-week intervals thereafter (on Day 1 of every odd-numbered Cycle of 28-days) through 15 Cycles and every 3 Cycles thereafter until disease progression or up to end of the study (approximately up to 69 months)
Population: ITT Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhered to the assigned dose.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
percentage of participants | 45.5 [34.8 to 56.5] | 57.3 [46.1 to 67.9]

2. Secondary Outcome: Confirmed Objective Response Rate (ORR) as Assessed by Independent Review Committee (IRC)
Description: ORR assessed by the IRC, was defined as the percentage of the participants with CR or PR according to RECIST v1.1 (confirmed ≥4 weeks after initial response), after the initiation of study treatment. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in theSLD of target lesions, taking as reference the baseline sum diameters. The exact 2-sided 95% confidence interval was calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
percentage of participants | 51.8 [42.1 to 61.3] | 56.4 [46.6 to 65.8]

3. Secondary Outcome: Confirmed Intracranial Central Nervous System Objective Response Rate (CNS ORR) in Participants With Measurable Active Brain Metastases
Description: Confirmed intracranial CNS ORR was defined as the percentage of the participants with CR or PR in the intracranial CNS per modification of RECIST v1.1 as evaluated by IRC after the initiation of study drug. Confirmed responses were those that persisted on repeat imaging 4 weeks or more after initial response. CR for target lesion: disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis). CR for non-target lesion: disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Screening, at 8-week intervals thereafter (on Day 1 of every odd-numbered Cycle of 28-days) through 15 Cycles and every 3 Cycles thereafter until disease progression or approximately up to 29 months
Population: ITT Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhered to the assigned dose. Participants with measurable active brain metastases at Baseline were evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 19 | 15
percentage of participants | 47.4 [24.4 to 71.1] | 73.3 [44.9 to 92.2]

4. Secondary Outcome: Confirmed Intracranial Central Nervous System Objective Response Rate (CNS ORR) in Participants With Only Non-measurable Active Brain Metastases
Description: Confirmed intracranial CNS ORR is defined as the percentage of the participants with CR or PR in the intracranial CNS per modification of RECIST v1.1 as evaluated by IRC after the initiation of study drug. Confirmed responses were those that persisted on repeat imaging 4 weeks or more after initial response. CR for target lesion: disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis). CR for non-target lesion: disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the Baseline sum diameters.
Time Frame: as for outcome 3
Population: ITT Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhered to the assigned dose. Participants with only non-measurable active brain metastases at Baseline were evaluated for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 33 | 36
percentage of participants | 12.1 [3.4 to 28.2] | 16.7 [6.4 to 32.8]

5. Secondary Outcome: Intracranial CNS Progression Free Survival (PFS) in Participants With Active Brain Metastases
Description: Intracranial CNS PFS as evaluated by IRC is defined as the time interval from the date of the first dose of the study drug until the first date at which intracranial CNS disease progression, an increase of 20% or more in the sum of diameters of intracranial CNS target lesions, unequivocal progression of non-target lesions, or the appearance of new lesions in the intracranial CNS, was objectively documented by a scan, or death due to any cause, whichever occurred first. The analysis was based on the Kaplan-Meier (KM) Estimates.
Time Frame: as for outcome 3
Population: ITT Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhered to the assigned dose. Participants with active brain metastases whether it was measurable or non-measurable at baseline were evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 52 | 51
months | 12.8 [9.0 to 18.4] | 12.8 [9.1 to 21.1]

6. Secondary Outcome: Time to Response
Description: Time to response was defined as the time interval from the date of the first dose of the study drug until the initial observation of CR or PR for participants with confirmed CR/PR. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the Baseline sum diameters.
Time Frame: Up to approximately 69 months
Population: ITT Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhered to the assigned dose. Participants who had confirmed CR or PR were evaluable for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 51 | 63
months | 1.8 [1.7 to 11.1] | 1.9 [1.0 to 35.0]

7. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time interval from the time that the measurement criteria are first met for CR/PR (whichever is first recorded) until the first date that the progressive disease is objectively documented or death. Patients without progressive disease or death were censored at the last valid response assessment. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. The analysis was based on the Kaplan-Meier (KM) Estimates.
Time Frame: Up to approximately 69 months
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 51 | 63
months | 12.0 [9.2 to 19.4] | 13.8 [10.8 to 17.6]

8. Secondary Outcome: Time on Treatment
Description: Time on treatment was defined as the time from the first to the last dose of study drug. For participants who have not discontinued, time on treatment was censored as of the last dose of the study drug.
Time Frame: Up to approximately 69 months
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: days
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 109 | 110
days | 402.0 [1 to 1882] | 522.0 [2 to 2030]

9. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of randomized participants who were confirmed to have achieved CR or PR or have a best overall response as stable disease (SD) for 6 weeks or more after initiation of the study drug. CR for target lesion: disappearance of all extranodal lesions and all pathological lymph nodes must have decreased to <10 mm in short axis. CR for non-target lesion: Disappearance of all extranodal non-target lesions, all lymph nodes must be non-pathological in size (<10mm short axis) and norrmalization of tumor marker level. PR: at least a 30% decrease in the SLD of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
percentage of participants | 81.3 [72.8 to 88.0] | 86.4 [78.5 to 92.2]

10. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time interval from the date of the first dose of the study treatment until the first date at which disease progression is objectively documented, or death due to any cause, whichever occurs first. Disease progression for target lesion: SLD increased by at least 20% from the smallest value on study (including Baseline, if that is the smallest) and SLD must also demonstrate an absolute increase of at least 5 mm or development of any new lesion. Disease progression for non-target lesion: Unequivocal progression of existing non-target lesions. (Subjective judgment by experienced reader). The analysis was based on the Kaplan-Meier (KM) Estimates.
Time Frame: Up to approximately 69 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
months | 9.2 [7.4 to 11.1] | 15.6 [11.1 to 18.5]

11. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time interval from the date of the first dose of the study treatment until death due to any cause. Intracranial OS was calculated by Kaplan-Meier estimation.
Time Frame: Up to approximately 69 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
months | 25.9 [18.2 to 45.8] | 40.6 [32.5 to NA] — Upper limit of 95% confidence interval was not estimable due to low number of participants with event.

12. Secondary Outcome: Number of Participants Who Had at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE was defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug up to 30 days following the last dose of study drug (approximately up to 69 months)
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 109 | 110
participants | 109 | 110

13. Secondary Outcome: Pre-dose Brigatinib Plasma Concentration
Time Frame: Day 1 Cycles 2, 3, 4 and 5 (each Cycle of 28-days) pre-dose
Population: ITT Population included all participants who were randomized to each regimen regardless of whether they received study drug or adhered to the assigned dose. Here, number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
ng/ml
  Cycle 2: number analyzed (Participants) | 101 | 97
  Cycle 2 | 295.2 (252.0) | 520.0 (321.9)
  Cycle 3: number analyzed (Participants) | 91 | 92
  Cycle 3 | 263.9 (238.9) | 537.0 (360.3)
  Cycle 4: number analyzed (Participants) | 80 | 87
  Cycle 4 | 236.1 (188.0) | 564.7 (415.0)
  Cycle 5: number analyzed (Participants) | 80 | 79
  Cycle 5 | 256.4 (282.3) | 579.7 (396.7)

14. Secondary Outcome: Patient-reported Symptoms Global Health Status/Quality of Life (QoL) Scores
Description: Patient-reported symptoms global health status/quality of life (QoL) scores were based on questions 29 and 30 of the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-C30 (QLQ-C30). The first 28 questions used 4-point scale (1=not at all,2=a little,3=quite a bit,4=very much) for evaluating 5 functional scales (physical, role, cognitive, emotional, and social functioning); 3 symptom scales (fatigue, pain, and nausea/vomiting); and last 2 questions on global health status/QoL scale are coded on 7-point scale (1=very poor to 7=excellent). Six single-item scales also are included (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Raw scores for multi-item scales and single-item measures was linearly transformed to obtain the score ranging from 0 to 100, where higher score represents a higher ("better") level of functioning.
Time Frame: Baseline and at each 28-day cycle up to end of the study (up to approximately 69 months)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
Number analyzed (Participants) | 112 | 110
unit on a scale
  Baseline: number analyzed (Participants) | 108 | 108
  Baseline | 52.39 (27.42) | 58.49 (23.40)
  Cycle 2: number analyzed (Participants) | 101 | 97
  Cycle 2 | 64.19 (20.73) | 65.72 (19.54)
  Cycle 3: number analyzed (Participants) | 91 | 91
  Cycle 3 | 65.57 (24.06) | 68.50 (20.52)
  Cycle 4: number analyzed (Participants) | 84 | 89
  Cycle 4 | 69.44 (20.59) | 66.95 (20.89)
  Cycle 5: number analyzed (Participants) | 82 | 85
  Cycle 5 | 70.12 (20.28) | 71.86 (17.63)
  Cycle 6: number analyzed (Participants) | 79 | 82
  Cycle 6 | 70.15 (20.18) | 71.24 (18.66)
  Cycle 7: number analyzed (Participants) | 77 | 80
  Cycle 7 | 67.42 (20.29) | 70.21 (21.66)
  Cycle 8: number analyzed (Participants) | 73 | 78
  Cycle 8 | 67.24 (22.79) | 69.87 (20.42)
  Cycle 9: number analyzed (Participants) | 70 | 75
  Cycle 9 | 68.45 (22.61) | 68.67 (21.35)
  Cycle 10: number analyzed (Participants) | 65 | 70
  Cycle 10 | 71.79 (20.61) | 67.98 (23.25)
  Cycle 11: number analyzed (Participants) | 61 | 70
  Cycle 11 | 72.54 (19.56) | 68.45 (21.37)
  Cycle 12: number analyzed (Participants) | 61 | 65
  Cycle 12 | 68.03 (23.08) | 70.51 (21.35)
  Cycle 13: number analyzed (Participants) | 58 | 64
  Cycle 13 | 70.11 (19.93) | 72.79 (19.20)
  Cycle 14: number analyzed (Participants) | 55 | 57
  Cycle 14 | 69.55 (20.04) | 70.76 (19.42)
  Cycle 15: number analyzed (Participants) | 54 | 58
  Cycle 15 | 70.06 (21.08) | 70.83 (20.66)
  Cycle 16: number analyzed (Participants) | 50 | 58
  Cycle 16 | 68.17 (22.94) | 72.27 (18.36)
  Cycle 17: number analyzed (Participants) | 48 | 61
  Cycle 17 | 73.61 (18.78) | 69.81 (20.36)
  Cycle 18: number analyzed (Participants) | 43 | 58
  Cycle 18 | 67.64 (22.80) | 71.55 (17.94)
  Cycle 19: number analyzed (Participants) | 43 | 55
  Cycle 19 | 69.57 (23.14) | 72.12 (20.49)
  Cycle 20: number analyzed (Participants) | 40 | 52
  Cycle 20 | 66.04 (24.05) | 72.76 (18.53)
  Cycle 21: number analyzed (Participants) | 39 | 50
  Cycle 21 | 69.23 (22.87) | 69.83 (19.04)
  Cycle 22: number analyzed (Participants) | 36 | 46
  Cycle 22 | 72.69 (21.70) | 71.20 (18.90)
  Cycle 23: number analyzed (Participants) | 35 | 47
  Cycle 23 | 72.38 (21.93) | 71.10 (20.10)
  Cycle 24: number analyzed (Participants) | 32 | 42
  Cycle 24 | 72.66 (19.66) | 71.43 (15.74)
  Cycle 25: number analyzed (Participants) | 34 | 39
  Cycle 25 | 71.57 (21.72) | 70.09 (19.38)
  Cycle 26: number analyzed (Participants) | 32 | 36
  Cycle 26 | 71.88 (22.28) | 69.68 (20.43)
  Cycle 27: number analyzed (Participants) | 33 | 36
  Cycle 27 | 71.46 (20.94) | 70.83 (21.96)
  Cycle 28: number analyzed (Participants) | 31 | 37
  Cycle 28 | 71.24 (22.24) | 69.59 (20.24)
  Cycle 29: number analyzed (Participants) | 30 | 37
  Cycle 29 | 70.00 (21.73) | 71.17 (22.27)
  Cycle 30: number analyzed (Participants) | 29 | 34
  Cycle 30 | 69.25 (21.72) | 70.83 (18.03)
  Cycle 31: number analyzed (Participants) | 26 | 33
  Cycle 31 | 75.64 (17.63) | 69.95 (18.15)
  Cycle 32: number analyzed (Participants) | 25 | 31
  Cycle 32 | 73.00 (20.02) | 70.97 (20.28)
  Cycle 33: number analyzed (Participants) | 25 | 32
  Cycle 33 | 71.67 (20.41) | 70.31 (20.84)
  Cycle 34: number analyzed (Participants) | 21 | 31
  Cycle 34 | 72.62 (20.61) | 69.62 (20.70)
  Cycle 35: number analyzed (Participants) | 21 | 31
  Cycle 35 | 72.22 (18.88) | 66.67 (22.97)
  Cycle 36: number analyzed (Participants) | 20 | 30
  Cycle 36 | 68.33 (22.72) | 71.67 (19.89)
  Cycle 37: number analyzed (Participants) | 20 | 30
  Cycle 37 | 73.33 (19.42) | 72.50 (19.47)
  Cycle 38: number analyzed (Participants) | 18 | 29
  Cycle 38 | 68.98 (22.10) | 72.99 (17.49)
  Cycle 39: number analyzed (Participants) | 17 | 26
  Cycle 39 | 68.63 (25.09) | 73.72 (19.96)
  Cycle 40: number analyzed (Participants) | 17 | 26
  Cycle 40 | 71.57 (24.13) | 69.87 (23.10)
  Cycle 41: number analyzed (Participants) | 17 | 26
  Cycle 41 | 72.55 (21.20) | 68.27 (22.98)
  Cycle 42: number analyzed (Participants) | 17 | 24
  Cycle 42 | 72.06 (21.84) | 72.57 (20.78)
  Cycle 43: number analyzed (Participants) | 17 | 23
  Cycle 43 | 67.65 (24.63) | 71.01 (22.17)
  Cycle 44: number analyzed (Participants) | 17 | 22
  Cycle 44 | 72.55 (20.57) | 73.48 (19.35)
  Cycle 45: number analyzed (Participants) | 14 | 22
  Cycle 45 | 66.67 (19.88) | 72.35 (22.03)
  Cycle 46: number analyzed (Participants) | 15 | 22
  Cycle 46 | 70.56 (19.12) | 71.59 (20.52)
  Cycle 47: number analyzed (Participants) | 14 | 21
  Cycle 47 | 60.12 (25.36) | 73.02 (19.88)
  Cycle 48: number analyzed (Participants) | 13 | 21
  Cycle 48 | 65.38 (20.93) | 74.60 (19.80)
  Cycle 49: number analyzed (Participants) | 13 | 20
  Cycle 49 | 57.69 (24.88) | 71.67 (22.69)
  Cycle 50: number analyzed (Participants) | 13 | 20
  Cycle 50 | 61.54 (26.47) | 70.00 (24.54)
  Cycle 51: number analyzed (Participants) | 12 | 21
  Cycle 51 | 63.19 (23.96) | 69.05 (22.69)
  Cycle 52: number analyzed (Participants) | 12 | 21
  Cycle 52 | 56.94 (22.71) | 72.22 (22.26)
  Cycle 53: number analyzed (Participants) | 12 | 20
  Cycle 53 | 61.11 (21.42) | 70.83 (23.02)
  Cycle 54: number analyzed (Participants) | 12 | 19
  Cycle 54 | 61.81 (25.24) | 71.49 (20.47)
  Cycle 55: number analyzed (Participants) | 10 | 19
  Cycle 55 | 63.33 (26.12) | 72.37 (20.42)
  Cycle 56: number analyzed (Participants) | 9 | 18
  Cycle 56 | 63.89 (23.94) | 73.61 (19.23)
  Cycle 57: number analyzed (Participants) | 10 | 17
  Cycle 57 | 65.00 (19.95) | 73.53 (19.37)
  Cycle 58: number analyzed (Participants) | 10 | 14
  Cycle 58 | 65.00 (25.09) | 70.83 (20.61)
  Cycle 59: number analyzed (Participants) | 9 | 14
  Cycle 59 | 64.81 (25.27) | 71.43 (19.81)
  Cycle 60: number analyzed (Participants) | 8 | 9
  Cycle 60 | 70.83 (27.82) | 73.15 (19.44)
  Cycle 61: number analyzed (Participants) | 7 | 8
  Cycle 61 | 71.43 (28.41) | 78.13 (19.89)
  Cycle 62: number analyzed (Participants) | 5 | 7
  Cycle 62 | 66.67 (23.57) | 79.76 (15.85)
  Cycle 63: number analyzed (Participants) | 4 | 7
  Cycle 63 | 58.33 (31.91) | 78.57 (17.91)
  Cycle 64: number analyzed (Participants) | 3 | 7
  Cycle 64 | 61.11 (34.69) | 77.38 (20.81)
  Cycle 65: number analyzed (Participants) | 2 | 6
  Cycle 65 | 75.00 (35.36) | 76.39 (22.62)
  Cycle 66: number analyzed (Participants) | 2 | 4
  Cycle 66 | 75.00 (35.36) | 77.08 (31.46)
  Cycle 67: number analyzed (Participants) | 2 | 1
  Cycle 67 | 75.00 (35.36) | 41.67 (NA) — Standard deviation (SD) was not evaluable for 1 participant.
  Cycle 68: number analyzed (Participants) | 0 | 1
  Cycle 68 |  | 41.67 (NA) — SD was not evaluable for 1 participant.
  Cycle 69: number analyzed (Participants) | 0 | 1
  Cycle 69 |  | 58.33 (NA) — SD was not evaluable for 1 participant.
  Cycle 70: number analyzed (Participants) | 0 | 1
  Cycle 70 |  | 41.67 (NA) — SD was not evaluable for 1 participant.
  Cycle 71: number analyzed (Participants) | 0 | 1
  Cycle 71 |  | 41.67 (NA) — SD was not evaluable for 1 participant.
  Cycle 72: number analyzed (Participants) | 0 | 1
  Cycle 72 |  | 75.00 (NA) — SD was not evaluable for 1 participant.
  End of Treatment: number analyzed (Participants) | 80 | 68
  End of Treatment | 52.29 (28.25) | 61.15 (23.15)
  Follow-Up 30 Days After Last Dose: number analyzed (Participants) | 43 | 45
  Follow-Up 30 Days After Last Dose | 61.05 (30.58) | 61.67 (23.33)

ADVERSE EVENTS:
Time Frame: All-cause Mortality: From first dose of study drug up to end of the study (approximately up to 69 months); Serious and Other Adverse Events: From first dose of study drug up to 30 days following the last dose of study drug (approximately up to 69 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Brigatinib 90 mg | Brigatinib 90 mg - 180 mg
All-Cause Mortality (participants affected / at risk) | 64/109 | 54/110
Serious Adverse Events (participants affected / at risk) | 58/109 | 69/110
Other Adverse Events (participants affected / at risk) | 108/109 | 105/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 90 mg (N=109) | Brigatinib 90 mg - 180 mg (N=110)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 8
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 13
Appendicitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 2 | 1
Atypical pneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 1 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Epilepsy (Nervous system disorders) | 3 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 4 | 1
Simple partial seizures (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Infusion site thrombosis (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Paraneoplastic dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Confusional state (Psychiatric disorders) | 2 | 2
Behcets syndrome (Vascular disorders) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bowens disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Tonic clonic movements (Nervous system disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal pain upper† (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Tooth socket haemorrhage (Gastrointestinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Hepatic function abnormal† (Hepatobiliary disorders) | 0 | 2
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Hypertension (Vascular disorders) | 0 | 1
Iliac artery stenosis (Vascular disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Device occlusion (Product Issues) | 1 | 1
Euthanasia (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brigatinib 90 mg (N=109) | Brigatinib 90 mg - 180 mg (N=110)
Nausea (Gastrointestinal disorders) | 47 | 55
Diarrhoea (Gastrointestinal disorders) | 34 | 51
Vomiting (Gastrointestinal disorders) | 44 | 39
Constipation (Gastrointestinal disorders) | 29 | 28
Abdominal pain (Gastrointestinal disorders) | 13 | 10
Dyspepsia (Gastrointestinal disorders) | 8 | 8
Stomatitis (Gastrointestinal disorders) | 5 | 10
Dry mouth (Gastrointestinal disorders) | 4 | 11
Headache (Nervous system disorders) | 39 | 44
Dizziness (Nervous system disorders) | 18 | 22
Paraesthesia (Nervous system disorders) | 13 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 10
Memory impairment (Nervous system disorders) | 4 | 11
Pyrexia (General disorders) | 23 | 11
Asthenia (General disorders) | 16 | 19
Oedema peripheral (General disorders) | 13 | 14
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 28
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 21
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 17
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 45
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Blood creatine phosphokinase increased (Investigations) | 24 | 41
Amylase increased (Investigations) | 16 | 20
Aspartate aminotransferase increased (Investigations) | 15 | 22
Lipase increased (Investigations) | 15 | 23
Alanine aminotransferase increased (Investigations) | 15 | 18
Blood lactate dehydrogenase increased (Investigations) | 3 | 10
Weight decreased (Investigations) | 8 | 7
Nasopharyngitis (Infections and infestations) | 15 | 15
Upper respiratory tract infection (Infections and infestations) | 13 | 10
Urinary tract infection (Infections and infestations) | 9 | 13
Rash (Skin and subcutaneous tissue disorders) | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 15
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 4
Decreased appetite (Metabolism and nutrition disorders) | 32 | 27
Hypertension (Vascular disorders) | 21 | 35
Insomnia (Psychiatric disorders) | 20 | 15
Vertigo (Ear and labyrinth disorders) | 3 | 13
Haematuria (Renal and urinary disorders) | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 11 | 13
Fatigue (General disorders) | 34 | 41
Influenza like illness (General disorders) | 8 | 9
Non-cardiac chest pain (General disorders) | 6 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6 | 4
Seizure (Nervous system disorders) | 4 | 11
Hypoaesthesia (Nervous system disorders) | 5 | 6
Cognitive disorder (Nervous system disorders) | 3 | 6
Tremor (Nervous system disorders) | 2 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Blood alkaline phosphatase increased (Investigations) | 7 | 6
Blood creatinine increased (Investigations) | 5 | 8
Electrocardiogram QT prolonged (Investigations) | 4 | 8
Pneumonia (Infections and infestations) | 3 | 15
Bronchitis (Infections and infestations) | 5 | 6
Sinusitis (Infections and infestations) | 3 | 8
Herpes zoster (Infections and infestations) | 1 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 9 | 14
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 8
Anxiety (Psychiatric disorders) | 3 | 11
Anaemia (Blood and lymphatic system disorders) | 8 | 8
Vision blurred (Eye disorders) | 7 | 9
Fall (Injury, poisoning and procedural complications) | 2 | 7
Palpitations (Cardiac disorders) | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2015-08-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT02094573/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT02094573/SAP_001.pdf